CLINICAL TRIAL: NCT04137731
Title: The Effect of Short Term Patient Outcomes With the Use of Interferential Current Therapy After Total Knee Arthroplasty
Brief Title: Use of Interferential Current (IFC) Therapy After Total Knee Arthroplasty
Acronym: IFC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Montefiore Medical Center (Other)
Collaborators: Ortho IFC LLC (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 2019-10138
Record Dates: First submitted 2019-10-22; First posted 2019-10-24 (Actual); Results first posted 2023-09-08 (Actual); Last update posted 2023-09-08 (Actual); Status verified 2023-09

CONDITIONS: Osteo Arthritis Knee
MeSH Terms: interventions — Electric Stimulation Therapy

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (2):
- IFC Treatment (Experimental): The IFC treatment will be used for 30 minutes, twice a day for two days after the total knee arthroplasty
  Interventions: Device: Interferential Current Therapy
- Placebo (Placebo Comparator): One set of device is programmed to be used as Placebo, the subject will feel the vibration but will not receive a therapeutic signal.
  Interventions: Device: Interferential Current Therapy

INTERVENTIONS:
Device: Interferential Current Therapy — IFC treatment after Total Knee Arthroplasty

SUMMARY:
Interferential Current Therapy (IFC) is a form of electrical therapy that utilizes two simultaneous low frequency electrical stimulation which when they cross interfere with one another resulting in an interference or beat frequency. This beat frequency provides a therapeutic area of relief by blocking painful stimuli at the area of interest. IFC is different from the other electrical treatment modalities used because the cancellation effect allows for establishment of the treatment area to be in the deeper tissues of the body, whereas other electrical modalities can only be used to treat superficial body parts that lie just under the skin.

The main objective of this proposed study is to assess the post-operative short term outcomes of the patients who receive IFC treatment during their post-total knee arthroplasty (TKA) surgery hospital stay. The implications of the study would be improved patient outcome which could result in shorter hospital stay, reduced use of opioid medication, decreased need for manipulation under anesthesia and reduced re-admission rate.

ELIGIBILITY:
Inclusion Criteria:Adult patients with knee osteoarthritis who have failed conservative therapy and undergoing elected TKA.

-

Exclusion Criteria:

i. <18 years old ii. Any patient with pacemaker or any electrical stimulator device iii. Patients without capacity to consent for the study iv. Patients not able to have local nerve block or spinal anesthesia v. Patients with prior chronic opioid use vi. Patients who are categorized to have 'Severe' fear and anxiety responses to pain, according to the Pain catastrophizing scale (PCS) survey.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2019-12-05 (Actual); Primary Completion 2022-08-15 (Actual); Study Completion 2022-08-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Zeynep Seref-Ferlengez, PhD, Principal Investigator — Albert Einstein College of Medicine; Sun Jin Kim, MD, Principal Investigator — Montefiore Medical Center
Locations (1):
- Montefiore Medical Center, The Bronx, New York, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: While forty-two (42) participants were consented, two of the consented participants never had surgery (one participant due to COVID-related restrictions and one participant on account of changing their mind) and thus were never enrolled/randomized into the study and thus 40 participants were considered to have been enrolled/randomized for purposes of analysis. Twenty into each arm/group
Period: Overall Study
Arm/Group | IFC Treatment | Placebo
Started | 20 | 20
Completed | 17 | 17
Not Completed | 3 | 3
Not completed — Surgery Cancellation | 1 | 2
Not completed — Withdrawal by Subject | 2 | 0
Not completed — Protocol Violation | 0 | 1

BASELINE CHARACTERISTICS:
Population: Baseline data provided for all 40 participants who were officially enrolled into the study. 20 participants per arm/group
Groups:
- Total: Total of all reporting groups
Arm/Group | IFC Treatment | Placebo | Total
Number analyzed (Participants) | 20 | 20 | 40
Age, Continuous [Mean (Standard Deviation); unit: Years] | 65.9 (10.5) | 65.2 (9.2) | 65.5 (9.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19 | 17 | 36
  Male | 1 | 3 | 4
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 7 | 7 | 14
  Not Hispanic or Latino | 6 | 10 | 16
  Unknown or Not Reported | 7 | 3 | 10
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 4 | 7 | 11
  White | 1 | 1 | 2
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 15 | 12 | 27
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 20 | 20 | 40

OUTCOME MEASURES:

1. Primary Outcome: Post-operative Opioid Pain Medication Usage
Description: Post-operative opioid pain medication usage was assessed by tabulating opioid use during the hospital stay after Total Knee Arthroplasty (TKA) as determined by median morphine milligram equivalents (MME).
Time Frame: 24 hours after surgery
Measure: Median (Inter-Quartile Range); unit: MME
Arm/Group | IFC Treatment | Placebo
Number analyzed (Participants) | 17 | 17
MME | 24.5 [15.0 to 34.0] | 15.0 [7.5 to 17]

2. Primary Outcome: Post-operative Opioid Pain Medication Usage
Description: Post-operative opioid pain medication usage was assessed by tabulating opioid use during the hospital stay after Total Knee Arthroplasty (TKA) as determined by median MME (morphine milligram equivalents).
Time Frame: 48 hours after surgery
Measure: Median (Inter-Quartile Range); unit: MME
Arm/Group | IFC Treatment | Placebo
Number analyzed (Participants) | 17 | 17
MME | 60.0 [48.8 to 70.0] | 60.0 [30.0 to 85.0]

3. Primary Outcome: Visual Pain Score (VAS)
Description: VAS asks a patient to mark a place on a scale that aligns with their level of pain smiley face 0=No pain - sad face 10=worst pain
Time Frame: 24 Hours after surgery
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | IFC Treatment | Placebo
Number analyzed (Participants) | 17 | 17
score on a scale | 6 [3 to 7] | 6 [4 to 8]

4. Primary Outcome: Visual Pain Score
Description: as for outcome 3
Time Frame: 48 Hours after surgery
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | IFC Treatment | Placebo
Number analyzed (Participants) | 17 | 17
score on a scale | 5.5 [3.75 to 7] | 6 [3.25 to 7]

ADVERSE EVENTS:
Time Frame: 3 months
Description: Adverse Event/Serious Adverse Events/Mortality was evaluated for the 17 participants in each arm/group who received the treatment or placebo
Arm/Group | IFC Treatment | Placebo
All-Cause Mortality (participants affected / at risk) | 0/17 | 0/17
Serious Adverse Events (participants affected / at risk) | 0/17 | 0/17
Other Adverse Events (participants affected / at risk) | 0/17 | 0/17

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-12-03): https://cdn.clinicaltrials.gov/large-docs/31/NCT04137731/Prot_SAP_000.pdf
  • Informed Consent Form (2019-12-03): https://cdn.clinicaltrials.gov/large-docs/31/NCT04137731/ICF_001.pdf